CLINICAL TRIAL: NCT00834197
Title: A Relative Bioavailability Study of 15 mg Mirtazapine Orally Disintegrating Tablets Under Non-Fasting Conditions
Brief Title: 15 mg Mirtazapine Orally Disintegrating Tablets, Non-Fasting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: R03-339
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Mirtazapine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Mirtazapine 15 mg (Orally Disintegrating) Tablets
- 2 (Active Comparator)
  Interventions: Drug: REMERON SolTab® 15 mg Orally Disintegrating Tablets

INTERVENTIONS:
Drug: Mirtazapine 15 mg (Orally Disintegrating) Tablets — 1 x 15 mg, single-dose non-fasting
  Arms: 1
Drug: REMERON SolTab® 15 mg Orally Disintegrating Tablets — 1 x 15 mg, single-dose non-fasting
  Arms: 2

SUMMARY:
This study will compare the relative bioavailability (rate and extent of absorption) of 15 mg Mirtazapine (Orally Disintegrating) Tablets manufactured by TEVA Pharmaceutical Industries, Ltd.; distributed by TEVA Pharmaceuticals USA with that of 15 mg REMERON SolTab® Orally Disintegrating Tablets manufactured for Organon Inc. by CIMA Labs Inc. following a single oral dose (1 x 15 mg) in healthy adult subjects under non-fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Screening Demographics: All subjects selected for this study will be healthy men or women 18 years of age or older at the time of dosing. The subject's body mass index (BMI) should be less than or equal to 30.
* Screening Procedures: Each subject will complete the screening process within 28 days prior to Period I dosing. Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed, and signed by each potential participant before fill implementation of screening procedures.
* Screening will include general observations, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature. The physical examination will include, but may not be limited to, an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems.
* The screening clinical laboratory will include:

  * Hematology: hematocrit, hemoglobin, WBC count with differential, RBC count, platelet count;
  * Clinical Chemistry: serum creatinine, BUN, glucose, AST(GOT), ALT(GPT), albumin, total bilirubin, total protein, and alkaline phosphatase;
  * HIV antibody, hepatitis B surface antigen, and hepatitis C antibody screens;
  * Urinalysis: by dipstick; full microscopic examination of dipstick positive; and
  * Urine Drug Screen: ethyl alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates and phencyclidine.
  * Serum Pregnancy Screen (female subjects only)
* If female and:

  * of childbearing potential, is practicing an acceptable barrier method of birth control for the duration of the study as judged by the investigator(s), such as condoms, sponge, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence; or
  * is postmenopausal for at least 1 year; or
  * is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

* Subjects with a recent history of drug or alcohol addiction or abuse.
* Subjects with the presence of a clinically significant disorder involving the cardiovascular, respiratory, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the clinical investigators).
* Subjects whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.
* Subjects demonstrating a positive hepatitis B surface antigen screen, hepatitis C antibody screen, or a reactive HIV antibody screen.
* Subjects demonstrating a positive pregnancy screen.
* Subjects who are currently breastfeeding.
* Subjects with a history of clinically significant allergies including drug allergies.
* Subjects with a history of allergic response(s) to mirtazapine or related drugs.
* Subjects with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators).
* Subjects who currently use of have used tobacco products within 90 days of Period I dosing.
* Subjects who have taken any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to Period I dosing.
* Subjects who report donating greater than 150 mL of blood within 28 days prior to Period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
* Subjects who have donated plasma (e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.
* Subjects who report receiving any investigational drug within 28 days prior to Period I dosing.
* Subjects who report taking any systemic prescription medication in the 14 days prior to Period I dosing.
* Subjects who report an intolerance of direct venipuncture.
* Subjects who report consuming an abnormal diet during the 28 days prior to Period I dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2003-07; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D. Carlson, Pharm. D., Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Test (Mirtazapine) First: 15 mg Mirtazapine Orally Disintegrating Tablets test product dosed in first period followed by 15 mg Remeron® SolTab™ Orally Disintegrating Tablets reference product dosed in the second period.
- Reference (Remeron®) First: 15 mg Remeron® SolTab™ Orally Disintegrating Tablets reference product dosed in first period followed by 15 mg Mirtazapine Orally Disintegrating Tablets test product dosed in the second period.
Period: First Intervention
Arm/Group | Test (Mirtazapine) First | Reference (Remeron®) First
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Washout of 14 Days
Arm/Group | Test (Mirtazapine) First | Reference (Remeron®) First
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Test (Mirtazapine) First | Reference (Remeron®) First
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test (Mirtazapine) First | Reference (Remeron®) First | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 10 | 12 | 22
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Black | 0 | 1 | 1
  White | 14 | 14 | 28
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration of Drug Substance in Plasma)
Description: Bioequivalence based on Cmax.
Time Frame: Blood samples collected over a 120 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Test (Mirtazapine): 15 mg Mirtazapine Orally Disintegrating Tablets test product dosed in either period.
- Reference (Remeron®): 15 mg Remeron® SolTab™ Orally Disintegrating Tablets reference product dosed in either period.
Arm/Group | Test (Mirtazapine) | Reference (Remeron®)
Number analyzed (Participants) | 32 | 32
pg/mL | 26345.06 (6917.71) | 25942.77 (5550.56)
Statistical Analysis 1: Comparison: Test (Mirtazapine) vs Reference (Remeron®); Test type: Non-Inferiority or Equivalence — The ANOVA model was utilized in comparing the effects between the test and reference products. Differences were declared statistically significant at the 5% level (p<0.05); Ratio of the T/R geometric mean x 100 = 100.59, 90% CI [95.76 to 105.65] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference and test product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on AUC0-t.
Time Frame: Blood samples collected over a 120 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Test (Mirtazapine) | Reference (Remeron®)
Number analyzed (Participants) | 32 | 32
pg*h/mL | 355137.72 (118663.09) | 359429 (112502.31)
Statistical Analysis 1: Comparison: Test (Mirtazapine) vs Reference (Remeron®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 98.17, 90% CI [94.82 to 101.65] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on AUC0-inf.
Time Frame: Blood samples collected over a 120 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Test (Mirtazapine) | Reference (Remeron®)
Number analyzed (Participants) | 32 | 32
pg*h/mL | 380545.78 (121850.49) | 385738.84 (118600.75)
Statistical Analysis 1: Comparison: Test (Mirtazapine) vs Reference (Remeron®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 98.25, 90% CI [95.22 to 101.39] — [estimate comment as in outcome 1, analysis 1]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.